CLINICAL TRIAL: NCT05966545
Title: Outcomes of Retained Posterior Segment Intraocular Foreign Body Extraction With Coexisting Cataract Via The Limbus or The Pars Plana Route
Brief Title: Extraction Routes of Intraocular Foreign Body
Acronym: IOFB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Abbas Abomesslam Ali Hashem, assistant lecturer, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZU-IRB#9040/24-10-24
Record Dates: First submitted 2023-07-21; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Intraocular Foreign Body
MeSH Terms: conditions — Eye Foreign Bodies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intraocular foreign body extraction via the limbus (Active Comparator): pars plana vitrectomy and intraocular foreign body removal via the limbus, after complete removal of adhesions around intraocular foreign body, then the foreign body will be grasped using basket forceps, and it will be brought to anterior chamber and then removed through limbal incision. The external earth magnet will be applied close to the limbus to prevent its slippage from the forceps if needed.
  Interventions: Procedure: pars plana vitrectomy and intraocular foreign body removal
- intraocular foreign body extraction via the pars plana route (Active Comparator): pars plana vitrectomy and intraocular foreign body removal via pars plana route, after complete removal of adhesions around intraocular foreign body, then IOFB will be grasped using basket forceps, and while the IOFB removed through the sclerotomy an external earth magnet will be applied close to the sclerotomy after enlargement the sclerotomy to prevent its slippage from the forceps and falling down onto the posterior pole if needed.
  Interventions: Procedure: pars plana vitrectomy and intraocular foreign body removal

INTERVENTIONS:
Procedure: pars plana vitrectomy and intraocular foreign body removal — removal of vitreous body and attachment to foreign body then extraction of foreign body

SUMMARY:
Intra ocular foreign body removal is indicated to avoid further many complications such as retinal detachment, endophthalmitis. The surgical approach for a posterior segment IOFB is pars plana vitrectomy and its extraction either through the pars plana. our study is to compare limbal route versus pars plana route for extraction of posterior segment IOFB associated with cataract as regard to safety and complications.

DETAILED DESCRIPTION:
Penetrating ocular injuries with retained posterior segment intraocular foreign body (IOFB) are relatively common and account for 17% to 41% of ocular injuries.

Intra ocular foreign body removal is indicated to avoid further many complications such as retinal detachment, endophthalmitis, retinal toxicity (secondary to chalcosis, siderosis) and sympathetic ophthalmia.

The surgical approach for a posterior segment IOFB is pars plana vitrectomy (PPV) and its extraction either through the pars plana or the limbus.

PPV and IOFB extraction through sclerotomy is the most commonly used approach. Most commonly retained posterior segment intra ocular foreign bodies (IOFB) are removed after enlarging one of the sclerotomy ports during pars plana vitrectomy. Intra operative complications reported during IOFB extraction were hypotony, vitreous hemorrhage, incarceration of the retina in the wound, IOFB slippage. Reported post-operative complications were glaucoma and retinal detachment. Incidence of post-operative RD was reported to range from 22% to 79% with poor visual outcomes in most cases PPV and IOFB extraction through the limbal route is an alternative approach to remove IOFB. Complications reported were less frequent and include microscopic hyphema and vitreous hemorrhage. The incidence of post-operative retinal detachment after IOFB extraction through limbus was reported to range from 7.15% to 27.7 % The limbal route for retained posterior segment IOFB extraction can offer the following advantages: it allows visually controlled delivery of the IOFB from the posterior pole to the limbal exit and it has no relation to the vitreous base, thus minimizing the risk of creating a peripheral retinal break during extraction of intraocular foreign body, in contrast to the hidden part behind the iris when using the pars plana route.

ELIGIBILITY:
Inclusion Criteria:

* Eyes with retained posterior segment intraocular foreign body associated with crystalline lens injury.
* Eyes with retained posterior segment intraocular foreign body associated with coexisting cataract.

Exclusion Criteria:

* Eyes with pre-operative retinal detachment
* Eyes with retained posterior segment IOFB with clear lens.
* Anterior segment IOFBs
* Severely damaged eyes with an initial visual acuity of no light perception where enucleation is the primary treatment
* Patients with severely traumatized cornea which can affect visualization during vitrectomy.
* Pseudophakic eyes.
* Eyes with endophthalmitis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
post-operative retinal detachment | 1, 3 and 6 months
  comparing incidence of post-operative retinal detachment after intraocular foreign body extraction via limbus versus pars plana route.

SECONDARY OUTCOMES:
post-operative best corrected visual acuity | 1, 3 and 6 months
  report post-operative best corrected visual acuity after intraocular foreign body extraction via limbus versus pars plana route.
associated intra operative and post-operative complications. | 1, 3 and 6 months
  report associated intra operative and post-operative complications

CONTACTS AND LOCATIONS:
Overall Officials: sherif A. Dabour, MD, Study Director — Zagazig University; Ahmad S. Khalil, MD, Study Director — Zagazig University
Locations (1):
- faculty of medicine, Zagazig university, Zagazig, Sharqia Province, Egypt

REFERENCES:
- [Background] Demircan N, Soylu M, Yagmur M, Akkaya H, Ozcan AA, Varinli I. Pars plana vitrectomy in ocular injury with intraocular foreign body. J Trauma. 2005 Nov;59(5):1216-8. doi: 10.1097/01.ta.0000196438.48182.ff. PMID 16385302
- [Background] Loporchio D, Mukkamala L, Gorukanti K, Zarbin M, Langer P, Bhagat N. Intraocular foreign bodies: A review. Surv Ophthalmol. 2016 Sep-Oct;61(5):582-96. doi: 10.1016/j.survophthal.2016.03.005. Epub 2016 Mar 17. PMID 26994871
- [Background] Wani VB, Al-Ajmi M, Thalib L, Azad RV, Abul M, Al-Ghanim M, Sabti K. Vitrectomy for posterior segment intraocular foreign bodies: visual results and prognostic factors. Retina. 2003 Oct;23(5):654-60. doi: 10.1097/00006982-200310000-00008. PMID 14574250
- [Background] Wickham L, Xing W, Bunce C, Sullivan P. Outcomes of surgery for posterior segment intraocular foreign bodies--a retrospective review of 17 years of clinical experience. Graefes Arch Clin Exp Ophthalmol. 2006 Dec;244(12):1620-6. doi: 10.1007/s00417-006-0359-6. PMID 16788826